CLINICAL TRIAL: NCT06614777
Title: Characterization of the Cytokine Profile and the Microbiome in Darier's Disease: Towards New Therapeutic Perspectives.
Brief Title: Characterization of the Cytokine Profile and the Microbiome in Darier's Disease
Acronym: DARKINBIOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/22/0509
Record Dates: First submitted 2024-08-26; First posted 2024-09-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Darier Disease
Keywords: Darier disease; cytokine profil,; microbiome; proteomic analysis; targeting therapy
MeSH Terms: conditions — Darier Disease

STUDY DESIGN:
Intervention Model Description: Interventional study, exploratory, prospective, descriptive, bicentric.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- investigation : biopsy and blood extraction (Experimental)
  Interventions: Procedure: skin biopsies and blood extraction

INTERVENTIONS:
Procedure: skin biopsies and blood extraction — Two 5 mm skin biopsies: lesional area and non-lesional area, on the trunk.
  * One blood sample (20 ml) to extract the plasma.
  * 15 successive tape-strippings in a lesional area.
  * Scans with two swabs: lesional area (preferably the trunk, 5 cm x 5 cm area) and non-lesional area.

SUMMARY:
Darier disease is a rare genetic skin disease caused by mutations in the ATP2A2 gene. Clinically, patients present with inflammatory and keratotic papules, sometimes erosive and oozing, predominating in seborrheic areas and folds. The lesions are very visible, causing itching and pain and a significant impairment of quality of life. Complications such as superinfections of the skin (bacterial and viral) are very common and sometimes severe. Therapeutically, treatments are mainly symptomatic and often of limited effectiveness, particularly on inflammation and pruritus. The main objective of this clinical study is to compare the microbiota of the epidermis of patients with Darier disease in non-lesional areas versus lesional areas , making it possible to identify bacteria/clusters of bacteria, but also to analyze the metabolic pathways of the microbiota associated with the microbial signature, until now not described. The secondary objectives envisaged are to study the correlation between this microbiotic profile and both the clinical characteristics of patients and the cytokine profile. The research will be performed on 40 patients aged 18 or over, suffering from moderate to severe Darier Disease. For each patient, several samples will be collected including biopsies, blood sample, swabbing and tape-stripping, on lesional and non-lesional areas.

DETAILED DESCRIPTION:
A study carried out in 75 patients showed the presence of Staphylococcus aureus in lesional skin in 68% of cases, this percentage being correlated with the affected surface and the severity of the disease. Histologically, there is a characteristic appearance of acantholytic dyskeratosis and the underlying dermis is the site of inflammation. On the physiopathological level, the mutations cause disturbances in calcium metabolism, causing a loss of cell adhesion and a disruption of keratinocyte differentiation. The mechanisms leading to inflammatory skin lesions and frequent superinfections are poorly understood and could be the consequence of the abnormality of the skin barrier, causing disturbances in the cytokine profile and the microbiota.

This has been shown in hereditary ichthyoses, another group of diseases with keratinization disorders, in which microbiota abnormalities and a TH17 cytokine profile have been demonstrated.

In Darier disease, a study published in 2023 also showed the presence of a TH17 profile in 6 patients.

In 2 patients, clinical improvement was also noted when using biotherapy targeting interleukin 17 or 23. Also in 2023, Amar et al. studied the skin microbiota of 14 patients and showed the presence of Staphylococcus aureus and Staphylococcus warneri in the inflammatory areas, the abundance of which correlated with the severity of the disease.

Our study will provide additional data to this recent work, by highlighting differential cytokine and microbiota signatures between the two skin areas studied, in order to validate our hypothesis of the involvement of cytokines and the microbiota in chronic skin inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over,
* MD (clinical diagnosis),
* MD moderate to severe,
* Person affiliated or beneficiary of a social security scheme,
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Other inflammatory dermatological diseases : atopic dermatitis, psoriasis and lichen planus,
* Skin superinfection (clinical diagnosis),
* Treatment with a biotherapy, in progress or in the 12 weeks preceding inclusion,
* Treatment with oral retinoids introduced in the 6 months preceding inclusion,
* Application of tacrolimus to the areas or to more than 30% of the body surface,
* Application of topical corticosteroids to the areas or to more than 30% of the body surface, within 2 weeks preceding inclusion,
* Oral corticosteroid therapy in the 2 weeks preceding inclusion,
* Application of topical retinoids to the areas in the 2 weeks prior to inclusion,
* Oral and/or topical antibiotic therapy in the 2 weeks preceding inclusion,
* Local antiseptic in the 2 weeks preceding inclusion,
* Local keratolytics on areas within 5 days preceding inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Comparison of microbiotic profiles (genomes of microorganisms) in lesional and non-lesional areas. | day 1
  Shotgun Metagenome Sequencing is used to learn what genomes are present in the sample

SECONDARY OUTCOMES:
Characterization qualitatively and quantitatively, at the epidermis level, the cytokine profile of patients (lesional skin, non-lesional skin) | Day 1
  This is a proteomic analysis of the cells of the sample
Correlation between the microbiotic profile observed on the epidermis (lesional skin) and the clinical characteristics of patients | Day 1
  Analysis of the symptoms of the patient and observation of the microbiotic profile to observe if microbiotic profile corresponds to clinical symptoms.
Comparison of the cytokine profile in the lesional area vs. non-lesional area, from the dermis (from a biopsy) of patients. | Day 1
  Analysis of the cytokines in each biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Mazereeuw-hautier, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, Centre Hospitalier Universitaire de Toulouse, France

IPD SHARING:
Plan to Share IPD: No